CLINICAL TRIAL: NCT06395454
Title: Procalcitonin as a Sepsis Biomarker in Guiding Antibiotics Treatment Duration in Ventilator Associated Pneumonia in Neuro-ICU: A Randomised Controlled Trial
Brief Title: Usage of Procalcitonin to Reduce Antibiotics Duration in VAP in Neurosurgical ICU
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Mohd Zulfakar Mazlan, MBBS, Associate Professor Dr, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USM/JEPeM/KK/24010018
Record Dates: First submitted 2024-04-24; First posted 2024-05-02 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Antibiotic Side Effect

STUDY DESIGN:
Intervention Model Description: In a parallel group design, participants are randomized to two groups (PCT guided versus Non PCT guided (standard of care).
  Each group receives a different intervention (e.g., pct vs crp, tw, blood culture, temperature and clinical).
  The groups are compared to assess the effectiveness of the interventions.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Procalcitonin guided antibiotics treatment duration (Experimental): Procalcitonin test in addition to standard care blood investigations
  Interventions: Diagnostic Test: Shorten antibiotics duration based on procalcitonin test levels
- Standard care guided antibiotics treatment duration (No Intervention)

INTERVENTIONS:
Diagnostic Test: Shorten antibiotics duration based on procalcitonin test levels — procalcitonin test will be taken on day 1 of recruitment as baseline, test done on day 5 will decide whether antibiotics will be withheld, followed by day 7 to determine rate of reinfection.
  Arms: Procalcitonin guided antibiotics treatment duration

SUMMARY:
Using Procalcitonin Tests to reduce antibiotics duration in Neurosurgical patients with Ventilated Associated Pneumonia

DETAILED DESCRIPTION:
Patients who are more than 18 years old who are admitted to Neurosurgical ICU will be recruited 48hours after ventilation if matches criteria for ventilator associated pneumonia. Patients will be randomised into 2 groups. first group will be procalcitonin guided in addition to conventionally guided sepsis assessment (TWC, CRP, body temperature). second group is only conventionally guided sepsis assessment. in procalcitonin guided group, blood sample will be taken on Day 1 of recruitment and day 5. On day 5 , the procalcitonin level will be compared to recommendations in PRORATA trial. If procalcitonin level is below the level to withhold antibiotics, recommendation will be made to the primary physician to off the antibiotics. Another Procalcitonin level will be repeated on Day 7 to rule out reinfection. This study aims to compare the duration of antibiotics and length of ICU stay among the 2 groups.

This study will fill up the gap among the lack of datas in neurosurgical patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to Neuro-ICU & Trauma ICU
* Patients aged >18 years old.
* Ventilation for >48 hours
* VAP and treated with antibiotics <24hours prior to inclusion in trial.
* Patient with arterial line or central line

Exclusion Criteria:

* Patients who are on antibiotics but not assumed or proven to have VAP
* Expected short ICU stay (<3 Days)
* Non-bacterial infections
* Long term antibiotic treatment (transplant or chemotherapy patients, endocarditis, osteomyelitis)
* Hospitalisation 48hours before enrolment
* Severe immunosuppression
* Pregnancy
* Primary team's decision to continue antibiotics for 14 days prior to trial
* DNAR or expected to die within 5 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Adults more than 18 years old
Enrollment: 48 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
To compare the duration of antibiotics between PCT versus Standard of care guided stopping antibiotic | 14 days
  compare the duration of antibiotics between 2 arms
To compare the length of ICU stay in between PCT versus Standard of care guided stopping antibiotic | 14 days
  compare the length of ICU stay in between 2 arms

SECONDARY OUTCOMES:
To compare 14 days mortality rate in between 2 arms | 14 days
  compare 14 days mortality rate in between 2 arms
To compare proportion of difficult to treat organisms (MRO) in between 2 arms | 14 days
  compare proportion of difficult to treat organisms (MRO) in between 2 arms
To compare the proportion of reinfection within 72 hours after stopping antibiotics | 14 days
  compare the proportion of reinfection within 72 hours after stopping antibiotics

CONTACTS AND LOCATIONS:
Overall Officials: Zulfakar Mazlan, Principal Investigator — Associated Professor Dr

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bonell A, Azarrafiy R, Huong VTL, Viet TL, Phu VD, Dat VQ, Wertheim H, van Doorn HR, Lewycka S, Nadjm B. A Systematic Review and Meta-analysis of Ventilator-associated Pneumonia in Adults in Asia: An Analysis of National Income Level on Incidence and Etiology. Clin Infect Dis. 2019 Jan 18;68(3):511-518. doi: 10.1093/cid/ciy543. PMID 29982303
- [Background] Papazian L, Klompas M, Luyt CE. Ventilator-associated pneumonia in adults: a narrative review. Intensive Care Med. 2020 May;46(5):888-906. doi: 10.1007/s00134-020-05980-0. Epub 2020 Mar 10. PMID 32157357
- [Background] Rhee C. Using Procalcitonin to Guide Antibiotic Therapy. Open Forum Infect Dis. 2016 Dec 7;4(1):ofw249. doi: 10.1093/ofid/ofw249. eCollection 2017 Winter. PMID 28480245
- [Background] Brunkhorst FM, Wegscheider K, Forycki ZF, Brunkhorst R. Procalcitonin for early diagnosis and differentiation of SIRS, sepsis, severe sepsis, and septic shock. Intensive Care Med. 2000 Mar;26 Suppl 2:S148-52. doi: 10.1007/BF02900728. PMID 18470710
- [Background] Schroeder S, Hochreiter M, Koehler T, Schweiger AM, Bein B, Keck FS, von Spiegel T. Procalcitonin (PCT)-guided algorithm reduces length of antibiotic treatment in surgical intensive care patients with severe sepsis: results of a prospective randomized study. Langenbecks Arch Surg. 2009 Mar;394(2):221-6. doi: 10.1007/s00423-008-0432-1. Epub 2008 Nov 26. PMID 19034493
- [Background] Z Mazlan M, A H Ismail M, Ali S, Salmuna ZN, Wan Muhd Shukeri WF, Omar M. Efficacy and safety of the point-of-care procalcitonin test for determining the antibiotic treatment duration in patients with ventilator-associated pneumonia in the intensive care unit: a randomised controlled trial. Anaesthesiol Intensive Ther. 2021;53(3):207-214. doi: 10.5114/ait.2021.104300. PMID 34006044
- [Background] Bouadma L, Luyt CE, Tubach F, Cracco C, Alvarez A, Schwebel C, Schortgen F, Lasocki S, Veber B, Dehoux M, Bernard M, Pasquet B, Regnier B, Brun-Buisson C, Chastre J, Wolff M; PRORATA trial group. Use of procalcitonin to reduce patients' exposure to antibiotics in intensive care units (PRORATA trial): a multicentre randomised controlled trial. Lancet. 2010 Feb 6;375(9713):463-74. doi: 10.1016/S0140-6736(09)61879-1. Epub 2010 Jan 25. PMID 20097417
- [Background] Vishalashi SG, Gupta P, Verma PK. Serum Procalcitonin as a Biomarker to Determine the Duration of Antibiotic Therapy in Adult Patients with Sepsis and Septic Shock in Intensive Care Units: A Prospective Study. Indian J Crit Care Med. 2021 May;25(5):507-511. doi: 10.5005/jp-journals-10071-23802. PMID 34177168
- [Background] Najafi A, Khodadadian A, Sanatkar M, Shariat Moharari R, Etezadi F, Ahmadi A, Imani F, Khajavi MR. The Comparison of Procalcitonin Guidance Administer Antibiotics with Empiric Antibiotic Therapy in Critically Ill Patients Admitted in Intensive Care Unit. Acta Med Iran. 2015;53(9):562-7. PMID 26553084
- [Background] Christ-Crain M, Stolz D, Bingisser R, Muller C, Miedinger D, Huber PR, Zimmerli W, Harbarth S, Tamm M, Muller B. Procalcitonin guidance of antibiotic therapy in community-acquired pneumonia: a randomized trial. Am J Respir Crit Care Med. 2006 Jul 1;174(1):84-93. doi: 10.1164/rccm.200512-1922OC. Epub 2006 Apr 7. PMID 16603606
- [Background] Annane D, Maxime V, Faller JP, Mezher C, Clec'h C, Martel P, Gonzales H, Feissel M, Cohen Y, Capellier G, Gharbi M, Nardi O. Procalcitonin levels to guide antibiotic therapy in adults with non-microbiologically proven apparent severe sepsis: a randomised controlled trial. BMJ Open. 2013 Feb 14;3(2):e002186. doi: 10.1136/bmjopen-2012-002186. Print 2013. PMID 23418298
- [Background] Hochreiter M, Kohler T, Schweiger AM, Keck FS, Bein B, von Spiegel T, Schroeder S. Procalcitonin to guide duration of antibiotic therapy in intensive care patients: a randomized prospective controlled trial. Crit Care. 2009;13(3):R83. doi: 10.1186/cc7903. Epub 2009 Jun 3. PMID 19493352
- [Background] Schuetz P, Christ-Crain M, Muller B. Procalcitonin and other biomarkers to improve assessment and antibiotic stewardship in infections--hope for hype? Swiss Med Wkly. 2009 Jun 13;139(23-24):318-26. doi: 10.4414/smw.2009.12584. PMID 19529989
- [Background] Iankova I, Thompson-Leduc P, Kirson NY, Rice B, Hey J, Krause A, Schonfeld SA, DeBrase CR, Bozzette S, Schuetz P. Efficacy and Safety of Procalcitonin Guidance in Patients With Suspected or Confirmed Sepsis: A Systematic Review and Meta-Analysis. Crit Care Med. 2018 May;46(5):691-698. doi: 10.1097/CCM.0000000000002928. PMID 29271844
- [Background] Kibe S, Adams K, Barlow G. Diagnostic and prognostic biomarkers of sepsis in critical care. J Antimicrob Chemother. 2011 Apr;66 Suppl 2:ii33-40. doi: 10.1093/jac/dkq523. PMID 21398306
- [Background] Mazlan MZ, Ghazali AG, Omar M, Yaacob NM, Nik Mohamad NA, Hassan MH, Wan Muhd Shukeri WF. Predictors of Treatment Failure and Mortality among Patients with Septic Shock Treated with Meropenem in the Intensive Care Unit. Malays J Med Sci. 2024 Feb;31(1):76-90. doi: 10.21315/mjms2024.31.1.7. Epub 2024 Feb 28. PMID 38456106
- [Background] Nik Nurfazleen MZ, Mohamad Hasyizan H, Laila Ab M, Zeti Norfidiyati S, Kamaruddin I, Mahamarowi O, Mohd Zulfakar M. Clinical characteristics and factors associated with diagnoses of ventilator and non-ventilator associated pneumonia in Intensive care unit. Med J Malaysia. 2021 May;76(3):353-359. PMID 34031334